CLINICAL TRIAL: NCT05418764
Title: Effect of Validated Skills Simulation With the Miya Model on Operating Room Performance of Vaginal Hysterectomy
Brief Title: Effect of Validated Skills Simulation With the Miya Model
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00072056
Record Dates: First submitted 2022-06-09; First posted 2022-06-14 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-07

CONDITIONS: Vaginal Hysterectomy
Keywords: vaginal surgery techniques; gynecological procedures; mid-urethral slings (MUS); simulation training

STUDY DESIGN:
Intervention Model Description: Study participants will be residents at participating institutions who agree to participate in the study.
Who Masked: Outcomes Assessor
Masking Description: Participants will perform five hysterectomies on the Miya Model with a trainer who is a sub-PI at each institution, with each of these training sessions filmed and then scored by blinded experts - o Residents in the simulation arm will train until they reach a score of 27 on the modified Vagina Surgical Skills Index (VSSI)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants will receive standardized training by performing five hysterectomies on the Miya Model with a trainer who is a sub-PI at each Institution, with each of these training sessions filmed and then scored by blinded experts - Residents in the simulation arm will train until they reach a score of 27 on the modified Vagina Surgical Skills Index (VSSI)
  Interventions: Other: Miyamodel Training
- Control group (No Intervention): The training will be whatever is standard at their Institution

INTERVENTIONS:
Other: Miyamodel Training — standardized training by performing five hysterectomies on the Miyamodel with a trainer who is a sub-PI at each institution
  Arms: Intervention group

SUMMARY:
Simulation training with the Miya Model will improve Operating Room performance of Vaginal Hysterectomy (VH) in novice surgeons and this phase of the study is designed to test that.

DETAILED DESCRIPTION:
Vaginal Hysterectomy (VH) is the desired hysterectomy technique of The American College of Obstetricians and Gynecologists (ACOG) since it is associated with less morbidity, quicker recovery and lower costs than laparoscopic and abdominal hysterectomy. Despite its well documented advantages, numbers nationwide in the US are declining. Of all minimally invasive hysterectomy procedures, the vaginal approach has been the only one demonstrating a consistent decrease in use from 25% of cases in 1998 to 17% of cases in 2010. A large part of this is due to inadequate training for this technique. There currently is no standardized curriculum for teaching VH, and training varies widely between residency programs. It is widely held that simulation training for surgical procedures improves outcome, but there is a need to validate this for vaginal surgery training.

ELIGIBILITY:
Inclusion Criteria:

* residents at participating Institutions
* residents have performed ten or fewer vaginal hysterectomies

Exclusion Criteria:

* having had prior training dedicated to vaginal hysterectomy
* having performed eleven or more vaginal hysterectomies in the OR

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-12-27 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Vaginal Surgical Skills Index (VSSI) scores - Control Group | Month 2
  compare scores between the control and intervention group to see if the standardized simulation training improves OR performance - Range 0 - 40; higher score indicates better performance
Vaginal Surgical Skills Index (VSSI) scores - Intervention Group | Month 2
  compare scores between the control and intervention group to see if the standardized simulation training improves OR performance - Range 0 - 40; higher score indicates better performance

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Kammire, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No